CLINICAL TRIAL: NCT00991497
Title: A Randomised Controlled Trial to Compare the Outcome of Localised Varicosity Compression for 24 Hours and 5 Days After Foam Sclerotherapy to Truncal Varices
Brief Title: A Trial to Compare the Outcome of Localised Varicosity Compression for 24 Hours and 5 Days After Foam Sclerotherapy to Truncal Varices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gloucestershire Hospitals NHS Foundation Trust (Other)
Responsible Party: Jonothan J Earnshaw, Gloucetershire Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06/Q2005/128
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Varicose Veins
Keywords: varicose veins; foam sclerotherapy; compression bandaging; duration
MeSH Terms: conditions — Varicose Veins | interventions — Compression Bandages

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 24 hours compression bandaging (Active Comparator)
  Interventions: Device: Compression bandaging
- 5 days compression bandaging (Active Comparator)
  Interventions: Device: Compression bandaging

INTERVENTIONS:
Device: Compression bandaging — Cotton wool padding will then be placed over the treated vein and secured in place by crepe bandaging. An above-knee TED stocking will be applied on top of this.

SUMMARY:
The purpose of this study is to compare the results of foam treatment of varicose veins (foam sclerotherapy) in patients who wear compression bandages for 24 hours or 5 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Proven truncal venous incompetence (of >1 second duration) on venous duplex scanning. (Great saphenous vein (GSV), small saphenous vein (SSV), anterior accessory thigh vein (AATV) or other major tributary).
* Agreed preference for foam sclerotherapy treatment.
* Signed consent form agreeing to be part of the trial.

Exclusion Criteria:

* Total deep venous reflux.
* Known allergy to liquid sclerosant.
* Pregnancy or breast feeding.
* Arterial disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Change in Aberdeen Varicose Vein Score from time of treatment to 2 and 6 weeks after treatment | 2 and 6 weeks

SECONDARY OUTCOMES:
Change in Burford pain score from time of treatment to 2 and 6 weeks after treatment | 2 and 6 weeks
Change in SF-36 score from time of treatment to 6 weeks after treatment. | 6 weeks
Target vein occlusion rate on duplex imaging at 6 weeks | 6 weeks
Number and type of complications seen | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jonothan J Earnshaw, FRCS, MD, Principal Investigator — Gloucestershire Royal Hospital NHS Trust
Locations (1):
- Gloucestershire Royal Hospital NHS Trust, Gloucester, Gloucestershire, United Kingdom

REFERENCES:
- [Derived] O'Hare JL, Stephens J, Parkin D, Earnshaw JJ. Randomized clinical trial of different bandage regimens after foam sclerotherapy for varicose veins. Br J Surg. 2010 May;97(5):650-6. doi: 10.1002/bjs.6951. PMID 20306530